CLINICAL TRIAL: NCT06299176
Title: Phase 1 Feasibility and Safety of Whole Heart Radiotherapy for End-stage Heart Failure: First In-human Treatments
Brief Title: Whole Heart Radiotherapy for End-stage Heart Failure
Acronym: ESHF-WHRT
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Tarek Hijal, Dr. Tarek Hijal, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESHF-WHRT (2024-10362)
Record Dates: First submitted 2023-12-21; First posted 2024-03-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure NYHA Class III; Heart Failure NYHA Class IV; End-stage Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: radiation therapy; radiotherapy; radiation; heart failure; cardiac radioablation; left ventricle ejection fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: 6 participants with end-stage heart failure (NYHA 3 or 4, LVEF < 30%) with no other standard of care therapy options to receive whole heart radiation therapy.
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Whole Heart Radiation Therapy (Experimental): Whole heart radiotherapy, 5 Gy in 1 fraction
  Interventions: Other: Whole Heart Radiation Therapy

INTERVENTIONS:
Other: Whole Heart Radiation Therapy — Radiation to the whole heart in one treatment with a prescribed dose of 5 Gy.

SUMMARY:
End-stage heart failure (ESHF) causes recurrent hospitalizations, cardiac arrhythmias, and intolerance to standard HF therapies are common as the disease progresses. Management focuses on controlling symptoms, correcting precipitants, avoiding triggers, and improving quality-of-life. The combination of recent preclinical and clinical data suggests that localized cardiac RT is relatively safe and has positive conductive and anti-proliferative effects in the "sick" heart. In this Phase 1 study, the investigators aim to assess the feasibility and safety of 5 Gy whole heart radiotherapy in six (6) ESHF participants with limited options for further medical therapy to control their disease. The investigators hypothesize that 5 Gy whole heart radiotherapy can improve LVEF and decrease blood markers of heart failure and inflammation including B-type natriuretic peptide (BNP), C-reactive protein (CRP), and troponins, while also having a very tolerable side effect profile.

DETAILED DESCRIPTION:
HEART FAILURE Heart Failure (HF) is a heterogeneous syndrome manifested by vascular congestion and/or peripheral hypoperfusion in the setting of structural and/or functional cardiac abnormalities. Congestion commonly presents with dyspnea, reduced exercise tolerance, and edema while hypoperfusion results in end-organ dysfunction. HF is a major public health problem and because of its age-dependent increase in incidence and prevalence, it's one of the leading causes of death and hospitalization among the elderly. As a consequence of the worldwide increase in life expectancy, and due to improvements in the treatment of HF in recent years, the proportion of participants that reach an advanced phase of the disease, so-called ESHF, is steadily growing.

HF is characterized by impairment in cardiac structure and function which, in its advanced phases, results in decreased cardiac output (hypoperfusion) and/or fluid buildup (congestion). Initially cardiac output (CO) is maintained through the Frank-Starling mechanism with LV dilation and wall thickening. Eventually myocardial contractility declines and stroke volume (SV) decreases . A compensatory increase in heart rate (HR) may initially help maintain cardiac output, but this too will ultimately fail to preserve output. Currently, patients with HF are most often categorized as having heart failure with reduced (HFrEF; LVEF <40%), mid-range (HFmrEF; LVEF 40-49%) or preserved ejection fraction (HFpEF; LVEF ≥50%). The four classical hemodynamic profiles of heart failure can be categorized in a two-by-two matrix based on filling pressures (presence or absence of congestion) and perfusion status (adequate/inadequate). Furthermore, patients are classified by the New York Heart Association (NYHA) based on the presence or absence of symptoms during rest and physical activity (Figure 2). Patients with ESHF typically live in the NYHA Class III-IV and in a fine balance between the "wet and warm" (i.e. relatively preserved perfusion but congested) and "wet and cold" (i.e. low perfusion and congested) categories.

The two principal pathways mediating the pathophysiology of heart failure are the sympathetic nervous system (SNS) and the renin-angiotensin system (RAS). These systems are innately related, having the ability to further activate each other and ultimately resulting in a chronic state of increased effective circulating volume. Over time, myocardial alterations result in reduced responsiveness to these adaptive mechanisms, and thus a drop in cardiac output ensues. Not surprisingly the principal HF therapies target these pathways. The primary therapies have been comprised of the triad of ACE inhibitors (or angiotensin receptor blockers [ARB] if intolerant), beta-adrenoreceptor antagonists (beta-blockers), and mineralocorticoid receptor antagonists (MRAs) titrated to target doses. Unfortunately, in ESHF, medical optimization is often not tolerated because of worsening hypotension, hyperkalemia, and renal dysfunction. There is often a need to reduce the dose or eliminate these therapies which is a well-established marker of poor prognosis. Once diagnosed with ESHF focus turns towards defining the optimal therapeutic approach with options including orthotopic heart transplant (OHT), left ventricular assist device (LVAD) and/or palliation. Ultimately, a combination of these three strategies is often required.

Left ventricular ejection fraction (LVEF) is generally viewed as a clinically useful phenotypic marker indicative of underlying pathophysiological mechanisms and sensitivity to therapy.

End-stage heart failure (ESHF) manifests as severe and often relentless symptoms of dyspnea, fatigue, abdominal discomfort and ultimately cardiac cachexia with renal and hepatic dysfunction frequently further complicating the process. Recurrent hospitalizations, cardiac arrhythmias, and intolerance to standard HF therapies are common as the disease progresses. Management focuses on controlling symptoms, correcting precipitants, avoiding triggers, and improving quality-of-life (QOL).

RADIATION THERAPY Radiation therapy involves delivering high energy x-rays precisely to a target with minimal dose to the surrounding clinical tissues. Accuracy in radiation therapy requires effective patient immobilization, precise target localization, and highly conformed dosimetry and isotropic dose fall-off. Dose calculations involve algorithms that account for effects of tissue heterogeneities, and the linear accelerators that deliver the treatment are also equipped with multileaf collimators and have the ability of using multiple non-overlapping beams of radiation as well as intensity modulated radiation therapy to maximize accuracy of target dose deposition while minimizing surrounding organ dose.

Radiation therapy is used in many malignant and benign conditions with a variety of dose and fractionation schemes. For malignant diseases in the palliative setting, radiation therapy is delivered to painful or progressive sites of disease in a highly focused manner with significant benefit on controlling pain, local progression, and quality of life. Typical doses for these types of treatment vary and can be limited to 8 Gy in a single fraction. These treatments are tolerated extremely well by almost all patients with almost no side effects.

Radiation therapy (RT) is utilized half of all patients with a cancer diagnosis. RT is effective in reducing populations of highly proliferative cells, a common feature of malignant disease. RT is also used successfully to treat many non-malignant disorders, including hyperproliferative and inflammatory conditions. The RT doses required for these non-malignant disorders are often much smaller and carry a lighter burden of adverse effects. Recently, a number of human and murine studies indicate that in heart failure (HF), proliferating macrophages and fibroblasts are major mediators of collateral tissue injury and progressive disease. Strategies that ablate these highly proliferative precursors in preclinical models attenuate features of heart failure progression.

The use of high-dose stereotactic radiation therapy in patients with cardiac arrhythmias, specifically ventricular tachycardia (VT), has been shown to reduce arrhythmia burden in several human clinical trials and case series. In these studies, a single dose (25 Gy) of non-invasive electrophysiologically guided localized RT was safe, substantially reduced VT, improved left ventricular ejection fraction (LVEF) and improved quality of life (QOL) in 50-70% of patients with no other options for therapy. The initial hypothesis for this effect was that RT would create a scar, similar to how invasive catheter therapies are utilized to ablate arrhythmias. However, subsequent mechanistic studies suggest that rather than simply scarring the targeted tissue, RT stimulates physiologic changes including increased sodium channel (NaV1.5) and connexin-43 (Cx-43) expression, increasing conduction velocity within the heart. These physiologic changes were also seen outside of the 25Gy target areas, suggesting that smaller doses of radiation is sufficient to stimulate these effects. Retrospective analysis of the RT dosimetry from patients treated for VT demonstrated that 5 Gy was reflective of the approximate whole heart dose received outside of the targeted scar in these patients. A recent hypothesis postulated that 5 Gy may be sufficient to upregulate pro-conductive proteins and signaling pathways while attenuating cardiac remodeling via decreasing levels of macrophages and fibroblasts; the primary proliferative precursors to adverse cardiac remodeling in many models of cardiac injury. This was investigated in murine heart failure models, which demonstrated that 5 Gy of cardiac radiation delivered after injury attenuated adverse cardiac remodeling, improved LVEF, reduced fibrosis, and decreased proliferation of macrophages and fibroblasts.

HYPOTHESIS The combination of recent preclinical and clinical data suggests that localized cardiac RT is relatively safe and has positive conductive and anti-proliferative effects in the "sick" heart. In this Phase 1 study, the investigators aim to assess the feasibility and safety of 5 Gy whole heart radiotherapy in six (6) ESHF participants with limited options for further medical therapy to control their disease in a 3+3 study design. The investigators hypothesize that 5 Gy whole heart radiotherapy is a safe therapy with a limited side effect profile that may improve LVEF and decrease blood markers of heart failure and inflammation including B-type natriuretic peptide (BNP), C-reactive protein (CRP), troponins, lactate, and neturophil to lymphocyte ratio.

INTERIM REVIEW OF DATA, ESCALATION, AND DE-ESCALATION CRITERIA A data safety and monitoring board (DSMB) composed of two radiation oncologists and one cardiologists outside of the study team will review the data 30 days after the first 3 participants are treated. They will have the authority to stop the study based on the following dose-limiting toxicity (DLT) rule: all 3 patients with grade 3+ toxicity, or any grade 4+ toxicity classified as probably, or definitely related to the study intervention. Toxicities are based on CTCAE v5.0 definitions. Following this review, for the purpose of escalation and de-escalation, escalation-limiting toxicity (ELT) will be defined as any grade 3+ toxicity considered possibly, probably, or definitely related to the treatment intervention.

The following de-escalation, and escalation rules will be applied. There will be, at most, 4 dose levels. Escalation and de-escalation rules follow.

* Dose 1 (5 Gy) - starting dose based on rationale described in protocol
* Dose 0 (3 Gy) - de-escalation dose following 2 ELTs
* Dose 2 (7 Gy) - escalation dose 1 following no ELTs at Dose 1
* Dose 3 (9 Gy) - escalation dose 2 if no ELTs encountered at Dose 2

Following the treatment of 3 patients at dose level 1 (5 Gy), If one patient experiences a ELT, then 3 additional patients are enrolled at dose level 1 (5 Gy), for a maximum of 6 patients. If none of these patients experience a ELT then 3 patients would be enrolled at dose level 2 (7 Gy). If only one of those 6 patients experience a ELT, then the next 3 patients will be enrolled at dose level 2 (7 Gy).

The study continues in this fashion until no more than 1 of 6 patients treated at the highest dose level experience a ELT. At any dose level, if 2 patients experience a ELT, then dose de-escalation is to occur, with 6 total patients enrolled at that dose level.

PARTICIPANT TREATMENT SIMULATION Prior to radiation treatment planning, participants will be immobilized and a free-breathing CT simulation with 3 mm slice thickness will be performed. Respiratory correlated four-dimensional tomographic (4D-CT) images will be acquired to assess the extent of cardiac and respiratory motion. The average CT derived from 4D-CT images will be used for target and organ at risk (OAR) delineation as well as radiotherapy treatment planning.

RADIATION THERAPY TARGET VOLUMES The treatment target will be delineated using conventional radiotherapy definitions. The clinical target volume (CTV) will be defined on the simulation CT as the entire contour of the muscular heart excluding the pericardium. An ITV will be generated based on the motion seen on the 4D-CT, to encompass the combined respiratory and cardiac motion during free-breathing. A planning target volume (PTV) of up to 5 mm will be generated as a volumetric expansion from the ITV to account for uncertainties in planning and treatment delivery. Prior to creating a radiation treatment plan, organs-at-risk (OARs) including the spinal cord, stomach, liver, spleen, trachea, bronchi, lungs, and esophagus will be delineated.

TREATMENT PLAN, EVALUATION, AND QUALITY ASSURANCE Participants will be prescribed between 3Gy and 9 Gy in 1 fraction depending on which stage of escalation/de-escalation the trial is at. The plan will be normalized aiming for 95% coverage of the PTV volume by the 100% isodose. RT will be delivered with a 6 MV energy beam, using volumetric modulated arc therapy (VMAT) through partial arcs. Beam geometry will be optimized to avoid any defibrillator or pacemaker in place. Quality assurance (QA) for each treatment plan includes a group review of contours and plan by the radiation oncology, cardiology and medical physics study team members, as well as the standard departmental two-step plan verification prior to treatment and presentation at departmental QA rounds.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* End-stage heart failure with NYHA class 3 or 4,
* LVEF ≤ 30%
* NT-Pro-BNP ≥ 1500 pg/mL
* on maximum medical therapy with progressive symptoms/disease as defined by their primary cardiologist and ineligible for advanced therapies including left ventricular assist devices and heart transplant

Exclusion Criteria:

* previous RT in the treatment field that precludes further RT
* active connective tissue disease
* interstitial pulmonary fibrosis
* Participants who are unable to be positioned in a manner where treatment can be safely delivered

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute adverse events definitely or probably related to radiation therapy at 30 days as per CTCAE v 5.0 | 30 days
  Safety Endpoint

SECONDARY OUTCOMES:
Overall survival | 6 months
  Death from any cause after treatment
Hospital stays | 6 months
  length of hospitalization after treatment due to heart failure exacerbation
Subacute adverse events | 30-90 days after treatment
  Adverse events definitely or probably related to radiation therapy
Late adverse events | 90 days to 6 months after treatment
  Adverse events definitely or probably related to radiation therapy
Medication Changes - dose | 6 months
  changes in dose of medications following radiotherapy
Medication Changes - number | 6 months
  changes innumber of medications following radiotherapy
Quality of life KCCQ | day 0, 6 weeks, 12 weeks, 24 weeks
  quality of life based on questionnaire results following treatment
Quality of life - SF-36 | day 0, 6 weeks, 12 weeks, 24 weeks
  quality of life based on questionnaire results following treatment
Troponin changes | 2 weeks, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 1 year
  Changes in value of blood marker.
Lactate changes | 2 weeks, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 1 year
  Changes in value of blood marker.
Renal Function | 2 weeks, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 1 year
  Changes in value of blood marker.
Neutrophil-to-Lymphocyte Ratio | 2 weeks, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 1 year
  Changes in value of blood marker.
b-natrurietic peptide | 2 weeks, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 1 year
  Changes in value of blood marker.
Change in mean left ventricle ejection fraction | 6 weeks, 12 weeks, 24 weeks, 1 year
  Change in Left ventricle ejaction fraction as measured by transthoracic echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Gerard, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Tarek Hijal, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Martin L Bernier, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
no public sharing, will share anonymized data if necessary for other collaborative projects in future following REB review

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P. 2016 ESC Guidelines for the Diagnosis and Treatment of Acute and Chronic Heart Failure. Rev Esp Cardiol (Engl Ed). 2016 Dec;69(12):1167. doi: 10.1016/j.rec.2016.11.005. No abstract available. English, Spanish. PMID 27894487
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Kemp CD, Conte JV. The pathophysiology of heart failure. Cardiovasc Pathol. 2012 Sep-Oct;21(5):365-71. doi: 10.1016/j.carpath.2011.11.007. Epub 2012 Jan 5. PMID 22227365
- [Background] Nohria A, Tsang SW, Fang JC, Lewis EF, Jarcho JA, Mudge GH, Stevenson LW. Clinical assessment identifies hemodynamic profiles that predict outcomes in patients admitted with heart failure. J Am Coll Cardiol. 2003 May 21;41(10):1797-804. doi: 10.1016/s0735-1097(03)00309-7. PMID 12767667
- [Background] Srinivasan, S. and R. Kundu, Fluid Management in Cardiogenic Shock, in Rational Use of Intravenous Fluids in Critically Ill Patients, M.L.N.G. Malbrain, et al., Editors. 2024, Springer International Publishing: Cham. p. 315-328.
- [Background] Borlaug BA, Redfield MM. Diastolic and systolic heart failure are distinct phenotypes within the heart failure spectrum. Circulation. 2011 May 10;123(18):2006-13; discussion 2014. doi: 10.1161/CIRCULATIONAHA.110.954388. No abstract available. PMID 21555723
- [Background] Paulus WJ, Tschope C. A novel paradigm for heart failure with preserved ejection fraction: comorbidities drive myocardial dysfunction and remodeling through coronary microvascular endothelial inflammation. J Am Coll Cardiol. 2013 Jul 23;62(4):263-71. doi: 10.1016/j.jacc.2013.02.092. Epub 2013 May 15. PMID 23684677
- [Background] McMurray JJ. Clinical practice. Systolic heart failure. N Engl J Med. 2010 Jan 21;362(3):228-38. doi: 10.1056/NEJMcp0909392. No abstract available. PMID 20089973
- [Background] Triposkiadis F, Butler J, Abboud FM, Armstrong PW, Adamopoulos S, Atherton JJ, Backs J, Bauersachs J, Burkhoff D, Bonow RO, Chopra VK, de Boer RA, de Windt L, Hamdani N, Hasenfuss G, Heymans S, Hulot JS, Konstam M, Lee RT, Linke WA, Lunde IG, Lyon AR, Maack C, Mann DL, Mebazaa A, Mentz RJ, Nihoyannopoulos P, Papp Z, Parissis J, Pedrazzini T, Rosano G, Rouleau J, Seferovic PM, Shah AM, Starling RC, Tocchetti CG, Trochu JN, Thum T, Zannad F, Brutsaert DL, Segers VF, De Keulenaer GW. The continuous heart failure spectrum: moving beyond an ejection fraction classification. Eur Heart J. 2019 Jul 1;40(26):2155-2163. doi: 10.1093/eurheartj/ehz158. PMID 30957868
- [Background] Spencer K, Parrish R, Barton R, Henry A. Palliative radiotherapy. BMJ. 2018 Mar 23;360:k821. doi: 10.1136/bmj.k821. No abstract available. PMID 29572337
- [Background] Schaue D, McBride WH. Opportunities and challenges of radiotherapy for treating cancer. Nat Rev Clin Oncol. 2015 Sep;12(9):527-40. doi: 10.1038/nrclinonc.2015.120. Epub 2015 Jun 30. PMID 26122185
- [Background] Micke O, Seegenschmiedt MH; German Working Group on Radiotherapy in Germany. Consensus guidelines for radiation therapy of benign diseases: a multicenter approach in Germany. Int J Radiat Oncol Biol Phys. 2002 Feb 1;52(2):496-513. doi: 10.1016/s0360-3016(01)01814-4. PMID 11872298
- [Background] Rodel F, Fournier C, Wiedemann J, Merz F, Gaipl US, Frey B, Keilholz L, Seegenschmiedt MH, Rodel C, Hehlgans S. Basics of Radiation Biology When Treating Hyperproliferative Benign Diseases. Front Immunol. 2017 May 3;8:519. doi: 10.3389/fimmu.2017.00519. eCollection 2017. PMID 28515727
- [Background] Dick SA, Epelman S. Chronic Heart Failure and Inflammation: What Do We Really Know? Circ Res. 2016 Jun 24;119(1):159-76. doi: 10.1161/CIRCRESAHA.116.308030. PMID 27340274
- [Background] Lafuse WP, Wozniak DJ, Rajaram MVS. Role of Cardiac Macrophages on Cardiac Inflammation, Fibrosis and Tissue Repair. Cells. 2020 Dec 31;10(1):51. doi: 10.3390/cells10010051. PMID 33396359
- [Background] Prabhu SD, Frangogiannis NG. The Biological Basis for Cardiac Repair After Myocardial Infarction: From Inflammation to Fibrosis. Circ Res. 2016 Jun 24;119(1):91-112. doi: 10.1161/CIRCRESAHA.116.303577. PMID 27340270
- [Background] Rurik JG, Tombacz I, Yadegari A, Mendez Fernandez PO, Shewale SV, Li L, Kimura T, Soliman OY, Papp TE, Tam YK, Mui BL, Albelda SM, Pure E, June CH, Aghajanian H, Weissman D, Parhiz H, Epstein JA. CAR T cells produced in vivo to treat cardiac injury. Science. 2022 Jan 7;375(6576):91-96. doi: 10.1126/science.abm0594. Epub 2022 Jan 6. PMID 34990237
- [Background] Bajpai G, Bredemeyer A, Li W, Zaitsev K, Koenig AL, Lokshina I, Mohan J, Ivey B, Hsiao HM, Weinheimer C, Kovacs A, Epelman S, Artyomov M, Kreisel D, Lavine KJ. Tissue Resident CCR2- and CCR2+ Cardiac Macrophages Differentially Orchestrate Monocyte Recruitment and Fate Specification Following Myocardial Injury. Circ Res. 2019 Jan 18;124(2):263-278. doi: 10.1161/CIRCRESAHA.118.314028. PMID 30582448
- [Background] Pedersen LN, Valenzuela Ripoll C, Ozcan M, Guo Z, Lotfinaghsh A, Zhang S, Ng S, Weinheimer C, Nigro J, Kovacs A, Diab A, Klaas A, Grogan F, Cho Y, Ataran A, Luehmann H, Heck A, Kolb K, Strong L, Navara R, Walls GM, Hugo G, Samson P, Cooper D, Reynoso FJ, Schwarz JK, Moore K, Lavine K, Rentschler SL, Liu Y, Woodard PK, Robinson C, Cuculich PS, Bergom C, Javaheri A. Cardiac radiation improves ventricular function in mice and humans with cardiomyopathy. Med. 2023 Dec 8;4(12):928-943.e5. doi: 10.1016/j.medj.2023.10.006. Epub 2023 Nov 28. PMID 38029754
- [Background] Lydiard PGDip S, Blanck O, Hugo G, O'Brien R, Keall P. A Review of Cardiac Radioablation (CR) for Arrhythmias: Procedures, Technology, and Future Opportunities. Int J Radiat Oncol Biol Phys. 2021 Mar 1;109(3):783-800. doi: 10.1016/j.ijrobp.2020.10.036. Epub 2020 Nov 5. PMID 33160007
- [Background] Robinson CG, Samson PP, Moore KMS, Hugo GD, Knutson N, Mutic S, Goddu SM, Lang A, Cooper DH, Faddis M, Noheria A, Smith TW, Woodard PK, Gropler RJ, Hallahan DE, Rudy Y, Cuculich PS. Phase I/II Trial of Electrophysiology-Guided Noninvasive Cardiac Radioablation for Ventricular Tachycardia. Circulation. 2019 Jan 15;139(3):313-321. doi: 10.1161/CIRCULATIONAHA.118.038261. PMID 30586734
- [Background] Zhang DM, Navara R, Yin T, Szymanski J, Goldsztejn U, Kenkel C, Lang A, Mpoy C, Lipovsky CE, Qiao Y, Hicks S, Li G, Moore KMS, Bergom C, Rogers BE, Robinson CG, Cuculich PS, Schwarz JK, Rentschler SL. Cardiac radiotherapy induces electrical conduction reprogramming in the absence of transmural fibrosis. Nat Commun. 2021 Sep 24;12(1):5558. doi: 10.1038/s41467-021-25730-0. PMID 34561429
- [Background] Lavine KJ, Epelman S, Uchida K, Weber KJ, Nichols CG, Schilling JD, Ornitz DM, Randolph GJ, Mann DL. Distinct macrophage lineages contribute to disparate patterns of cardiac recovery and remodeling in the neonatal and adult heart. Proc Natl Acad Sci U S A. 2014 Nov 11;111(45):16029-34. doi: 10.1073/pnas.1406508111. Epub 2014 Oct 27. PMID 25349429
- [Background] Schilling JD, Machkovech HM, Kim AH, Schwendener R, Schaffer JE. Macrophages modulate cardiac function in lipotoxic cardiomyopathy. Am J Physiol Heart Circ Physiol. 2012 Dec 1;303(11):H1366-73. doi: 10.1152/ajpheart.00111.2012. Epub 2012 Oct 5. PMID 23042950
- [Background] Le Tourneau C, Lee JJ, Siu LL. Dose escalation methods in phase I cancer clinical trials. J Natl Cancer Inst. 2009 May 20;101(10):708-20. doi: 10.1093/jnci/djp079. Epub 2009 May 12. PMID 19436029
- [Background] Busija L, Pausenberger E, Haines TP, Haymes S, Buchbinder R, Osborne RH. Adult measures of general health and health-related quality of life: Medical Outcomes Study Short Form 36-Item (SF-36) and Short Form 12-Item (SF-12) Health Surveys, Nottingham Health Profile (NHP), Sickness Impact Profile (SIP), Medical Outcomes Study Short Form 6D (SF-6D), Health Utilities Index Mark 3 (HUI3), Quality of Well-Being Scale (QWB), and Assessment of Quality of Life (AQoL). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S383-412. doi: 10.1002/acr.20541. No abstract available. PMID 22588759
- [Background] Khajavi A, Moshki M, Minaee S, Vakilian F, Montazeri A, Hashemizadeh H. Chronic heart failure health-related quality of life questionnaire (CHFQOLQ-20): development and psychometric properties. BMC Cardiovasc Disord. 2023 Mar 29;23(1):165. doi: 10.1186/s12872-023-03197-9. PMID 36991337
- [Background] Timmerman R. A Story of Hypofractionation and the Table on the Wall. Int J Radiat Oncol Biol Phys. 2022 Jan 1;112(1):4-21. doi: 10.1016/j.ijrobp.2021.09.027. No abstract available. PMID 34919882
- [Background] Desai MY, Windecker S, Lancellotti P, Bax JJ, Griffin BP, Cahlon O, Johnston DR. Prevention, Diagnosis, and Management of Radiation-Associated Cardiac Disease: JACC Scientific Expert Panel. J Am Coll Cardiol. 2019 Aug 20;74(7):905-927. doi: 10.1016/j.jacc.2019.07.006. PMID 31416535